CLINICAL TRIAL: NCT02464176
Title: The Effects of Systemic Steroids on the Duration of a Psoas Compartment Block.
Brief Title: Systemic Steroids for Peripheral Nerve Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00032805
Record Dates: First submitted 2015-06-01; First posted 2015-06-08 (Estimated); Results first posted 2018-01-16 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-07

CONDITIONS: Osteoarthritis, Hip
Keywords: Arthroplasty, Hip, Replacement; Anesthesia, Local; Anesthesia Conduction; Bupivacaine; Dexamethasone; Preanesthetic Medications; Nerve Block; Lumbar Plexus Block; Analgesia; Glucocorticoids; Local Anesthetics
MeSH Terms: conditions — Osteoarthritis, Hip; Agnosia | interventions — Dexamethasone; dexamethasone 21-phosphate; Bupivacaine; Epinephrine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 4 mg dexamethasone group (Experimental): Following lumbar plexus nerve block administration using bupivacaine and epinephrine, 4 mg of systemic dexamethasone will be administered to this group intravenously. The volume given intravenously will be identical for all groups.
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine; Drug: Epinephrine; Procedure: Lumbar Plexus Nerve Block
- 8 mg dexamethasone group (Experimental): Following peripheral nerve block using bupivacaine and epinephrine administration, 8 mg of systemic dexamethasone will be administered to this group intravenously. The volume given intravenously will be identical for all groups.
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine; Drug: Epinephrine; Procedure: Lumbar Plexus Nerve Block
- Control Group (Placebo Comparator): Normal saline will be used as a placebo control group given at the same time and in the same manner as the experimental groups following peripheral nerve block administration. The volume given intravenously will be identical for all groups.
  Interventions: Drug: Bupivacaine; Drug: Epinephrine; Procedure: Lumbar Plexus Nerve Block; Drug: Saline

INTERVENTIONS:
Drug: Dexamethasone — A lumbar plexus nerve block will be performed for patients undergoing hip arthroplasty. A total of 25cc's of 0.25% bupivacaine with 1:400,000 epinephrine will be administered for postoperative analgesia. Surgical anesthesia will be provided either by an intrathecal spinal block or general anesthesia. Successful blockade will be assumed if the patient has a decrease or loss of pinprick sensation in the femoral nerve distribution, which innervates the anterior thigh. If no evidence of blockade is present, testing will occur again at 30 minutes post block. Testing will be performed with a 25 gauge Whitacre needle and once present the area of testing will be marked with a surgical marking pen so that repeat sensory testing can be undertaken at that same site over the course of the study. The subjects will then receive dexamethasone (4 or 8 mg) or placebo (saline) based on arm placement.
  Other Names: dexamethasone sodium phosphate injection
  Arms: 4 mg dexamethasone group; 8 mg dexamethasone group
Drug: Bupivacaine — Bupivacaine will be used in lumbar plexus nerve block mixture.
  Other Names: Bupivacaine Hydrochloride
Drug: Epinephrine — Epinephrine will be used in lumbar plexus nerve block mixture.
  Other Names: Adrenaline
Procedure: Lumbar Plexus Nerve Block — This is the procedure that will be performed.
Drug: Saline — Patients randomized to the placebo group will receive normal saline intravenously.
  Other Names: Normal saline, NaCl
  Arms: Control Group

SUMMARY:
This study will investigate the ability of systemic dexamethasone to prolong the sensory block duration for lumbar plexus nerve blockade.

DETAILED DESCRIPTION:
The purpose of this randomized, double-blinded, placebo-controlled trial is to examine the equivalency of two different doses of dexamethasone when given intravenously as an adjuvant medication for postoperative pain management. Specifically, this study will investigate the prolongation of time to recovery of sensation following a lumbar plexus block in patients undergoing total hip arthroplasties. The investigators hypothesize that dexamethasone will prolong the sensory block time when compared to placebo and that similar results will be obtained in the 4 mg arm when compared to the 8 mg arm. The primary end point will be time to sensory recovery in the femoral nerve cutaneous distribution (part of the lumbar plexus) as determined by pin-prick sensation assessment. Secondary endpoints will include, but are not be limited to: time to first opioid administration, total opioid consumption over 30 hours, and rest and incident verbal numerical pain scores at 6,12,18,24 and 30 hours post block placement.

ELIGIBILITY:
Inclusion Criteria: Primary elective total hip arthroplasty surgery

* must be a candidate for placement of a lumbar plexus block under anatomic landmark technique using electrical stimulation
* must give written informed consent for anesthesia
* must also be reliable and able to give accurate verbal pain scores postoperatively

Exclusion Criteria:

* contraindications to regional anesthesia including, allergy to amide local anesthetics, presence of peripheral neurologic dysfunction, pre-existing coagulopathy or infection in the area of interest will be excluded.
* insulin and non-insulin dependent diabetes mellitus
* preoperative use of systemic corticosteroids within 30 days of surgery
* chronic opioid use (defined as daily opioid dose of greater than 40 mg of oxycodone equivalents or any long-acting opioid)
* pregnancy
* failure to effectively place the lumbar plexus block.
* known prior adverse reaction to dexamethasone (for example: psychosis) or an allergy to dexamethasone

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daryl S Henshaw, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Turner JD, Dobson SW, Weller RS, Russell GB, Henshaw DS. Intravenous dexamethasone fails to prolong psoas compartment block when assessed by objective pinprick sensory testing: a prospective, randomised, dose-dependent, placebo-controlled equivalency trial. Br J Anaesth. 2018 Feb;120(2):308-316. doi: 10.1016/j.bja.2017.11.073. Epub 2017 Dec 1. PMID 29406180

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study run from June 2015 to January 2017 at Wake Forest Baptist Medical Center
Pre-assignment Details: Patients 18-90 years old undergoing primary elective total hip arthroplasty were eligible. Exclusion: contraindications to regional anaesthesia, peripheral neurologic dysfunction or neuropathy, diabetes mellitus, systemic corticosteroid use within 30-days of surgery, chronic opioid use, pregnancy, allergy or adverse reaction to dexamethasone.
Period: Overall Study
Arm/Group | 4 mg Dexamethasone Group | 8 mg Dexamethasone Group | Control Group
Started | 50 | 50 | 15
Completed | 50 | 50 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 4 mg Dexamethasone Group: Following lumbar plexus nerve block administration using bupivacaine and epinephrine, 4 mg of systemic dexamethasone will be administered to this group intravenously. The volume given intravenously will be identical for all groups.
  Dexamethasone: A lumbar plexus nerve block will be performed for patients undergoing hip arthroplasty. A total of 25cc's of 0.25% bupivacaine with 1:400,000 epinephrine will be administered for postoperative analgesia. Surgical anesthesia will be provided either by an intrathecal spinal block or general anesthesia. The block will be tested for block success. Testing will be performed with a 25 gauge Whitacre needle . The subjects will then receive dexamethasone (4 or 8 mg) or placebo (saline) based on arm placement.
  Bupivacaine: Bupivacaine will be used in lumbar plexus nerve block mixture.
  Epinephrine: Epinephrine will be used in lumbar plexus nerve block mixture.
  Lumbar Plexus Nerve Block: This is the procedure that will be performed.
- 8 mg Dexamethasone Group: Following peripheral nerve block using bupivacaine and epinephrine administration, 8 mg of systemic dexamethasone will be administered to this group intravenously. The volume given intravenously will be identical for all groups.
  Dexamethasone: A lumbar plexus nerve block will be performed for patients undergoing hip arthroplasty. A total of 25cc's of 0.25% bupivacaine with 1:400,000 epinephrine will be administered for postoperative analgesia. Surgical anesthesia will be provided either by an intrathecal spinal block or general anesthesia. The block will be tested for block success. Testing will be performed with a 25 gauge Whitacre needle . The subjects will then receive dexamethasone (4 or 8 mg) or placebo (saline) based on arm placement.
  Bupivacaine: Bupivacaine will be used in lumbar plexus nerve block mixture.
  Epinephrine: Epinephrine will be used in lumbar plexus nerve block mixture.
  Lumbar Plexus Nerve Block: This is the procedure that will be performed.
- Total: Total of all reporting groups
Arm/Group | 4 mg Dexamethasone Group | 8 mg Dexamethasone Group | Control Group | Total
Number analyzed (Participants) | 50 | 50 | 15 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 32 | 8 | 74
  >=65 years | 16 | 18 | 7 | 41
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [51 to 68] | 63 [56 to 71] | 66 [62 to 72] | 63 [57 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 27 | 5 | 52
  Male | 30 | 23 | 10 | 63
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 15 | 115
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 29.8 [25.5 to 36.1] | 29.3 [25.6 to 32.6] | 28.3 [22.7 to 34.2] | 29.3 [25.45 to 34.05]

OUTCOME MEASURES:

1. Primary Outcome: Duration of Sensory Blockade
Description: The primary outcome will be duration of sensory blockade in the distribution of the lumbar plexus as determined by pin-prick sensation as tested every two hours with pin-prick sensation.
Time Frame: 30 hours
Measure: Mean (Standard Deviation); unit: hours
Groups:
- 4 mg Dexamethasone Group: Following lumbar plexus nerve block administration using bupivacaine and epinephrine, 4 mg of systemic dexamethasone will be administered to this group intravenously. The volume given intravenously will be identical for all groups.
  Dexamethasone: A lumbar plexus nerve block will be performed for patients undergoing hip arthroplasty. A total of 25cc's of 0.25% bupivacaine with 1:400,000 epinephrine will be administered for postoperative analgesia. Surgical anesthesia will be provided either by an intrathecal spinal block or general anesthesia. Successful blockade will be assumed if the patient has a decrease or loss of pinprick sensation in the femoral nerve distribution, which innervates the anterior thigh. If no evidence of blockade is present, testing will occur again at 30 minutes post block. Testing will be performed with a 25 gauge Whitacre needle
- 8 mg Dexamethasone Group: Following peripheral nerve block using bupivacaine and epinephrine administration, 8 mg of systemic dexamethasone will be administered to this group intravenously. The volume given intravenously will be identical for all groups.
  Dexamethasone: A lumbar plexus nerve block will be performed for patients undergoing hip arthroplasty. A total of 25cc's of 0.25% bupivacaine with 1:400,000 epinephrine will be administered for postoperative analgesia. Surgical anesthesia will be provided either by an intrathecal spinal block or general anesthesia. Successful blockade will be assumed if the patient has a decrease or loss of pinprick sensation in the femoral nerve distribution, which innervates the anterior thigh. If no evidence of blockade is present, testing will occur again at 30 minutes post block. Testing will be performed with a 25 gauge Whitacre needle and once present the area of testing will be marked with a surgical marking pen so that repeat sensory testing can be undertaken
Arm/Group | 4 mg Dexamethasone Group | 8 mg Dexamethasone Group | Control Group
Number analyzed (Participants) | 50 | 50 | 15
hours | 18.5 (8) | 18.1 (7.1) | 19.6 (6.7)

2. Secondary Outcome: Time to First Analgesic Request
Description: Time (in minutes) will be recorded to first analgesic request following the block placement
Time Frame: 30 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | 4 mg Dexamethasone Group | 8 mg Dexamethasone Group | Control Group
Number analyzed (Participants) | 50 | 50 | 15
minutes | 474 [382 to 590] | 533 [415 to 716] | 432 [383 to 491]

3. Secondary Outcome: Total Opioid Consumption
Time Frame: 30 hours
Measure: Median (Inter-Quartile Range); unit: oxycodone mg equivalents
Arm/Group | 4 mg Dexamethasone Group | 8 mg Dexamethasone Group | Control Group
Number analyzed (Participants) | 50 | 50 | 15
oxycodone mg equivalents | 36.6 [25.0 to 55] | 30 [20 to 45] | 39.2 [30 to 63.3]

4. Secondary Outcome: Verbal Numeric Pain Score Comparisons
Description: This secondary outcome includes pain scores utilizing the verbal numeric pain score scale (0 to 11). Higher values indicate worse outcomes (higher pain scores). Lower values are better.
Time Frame: 24 hour
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | 4 mg Dexamethasone Group | 8 mg Dexamethasone Group | Control Group
Number analyzed (Participants) | 49 | 48 | 15
scores on a scale | 3 [1 to 4] | 2 [1 to 4] | 3 [2 to 5]

ADVERSE EVENTS:
Time Frame: Each participant was specifically monitored over a 30 hour time period while in the hospital and encouraged to report and adverse events while in the hospital or after while the study was being conducted.
Arm/Group | 4 mg Dexamethasone Group | 8 mg Dexamethasone Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/15
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes